CLINICAL TRIAL: NCT06789094
Title: Validating the Ain Shams Cognitive Assessment (ASCA) for Diagnosing Mild Cognitive Impairment and Dementia
Brief Title: Validating the Ain Shams Cognitive Assessment Tool
Acronym: ASCA
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doha Rasheedy, Professor of Geriatrics and Gerontology, Ain Shams University
Other Study IDs: FMASU R310/2024
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Mild Cognitive Impairment (MCI); Dementia
Keywords: Mild cognitive impairment; Dementia; cognitive assessment; Arabic cognitive assessment tools
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — Equipment and Supplies; Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Dementia: participants >60 years with Dementia diagnosed by DSM-5 criteria
  Interventions: Other: Ain Shams University Cognitive Assessment (ASCA) tool
- Mild cognitive impairment: participants >60 years with Mild cognitive impairment (MCI) diagnosed by DSM-5 criteria
  Interventions: Other: Ain Shams University Cognitive Assessment (ASCA) tool
- control: euthymic healthy community dwelling adult participants of various socioeconomic and educational status.
  Interventions: Other: Ain Shams University Cognitive Assessment (ASCA) tool

INTERVENTIONS:
Other: Ain Shams University Cognitive Assessment (ASCA) tool — The ASCA, developed at Ain Shams University, is a comprehensive tool designed for cognitive assessment in Egyptian population. It encompasses various tests to assess cognitive functions and cultural understanding. These include the Verbal Paired Associated Test, evaluating verbal learning, distractor interval, delayed recall, and word recognition. The Bender Gestalt assesses visual-motor skills and memory. Short-term and working memory are tested through Digit Forward and Digit Backward Span Length tasks. Set Shifting is measured using a modified Trail Making Test, adapted for illiterates. Additionally, tests for letter/lexical fluency, verbal fluency, language object naming, abstraction, and judgment offer further insights into cognitive abilities and cultural interpretation.
  Other Names: Patient Health Questionnaire 9; activity of daily living questionnaire

SUMMARY:
The diagnosis of cognitive impairment, including dementia and mild cognitive impairment (MCI), is crucial for timely intervention and management. Various screening tools are available for assessing cognitive function, among which the Mini-Mental State Examination (MMSE), the Addenbrooke's Cognitive Examination (ACE), and the Montreal Cognitive Assessment (MoCA) are widely used. However, the recently developed Ain Shams University Cognitive Assessment (ASCA) has shown promise in detecting early cognitive decline. This study aims to assess the performance of ASCA in diagnosing cognitive impairment against DSM5 criteria.

ELIGIBILITY:
Inclusion Criteria: older adult participants 60 years old and above who are native Arabic speakers

-

Exclusion Criteria:

* severe dementia, delirium, major mental disorders, aphasia, and those with severe visual or hearing impairment that interfere with the assessment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community dwelling elderly participants (caregivers of inpatients, attendants of primary care , elderly clubs and other community gatherings).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
ASCA cut off points | 4 months
  obtain cut-off scores for diagnosing mild cognitive impairment (MCI) and dementia using the Ain Shams Cognitive Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided